CLINICAL TRIAL: NCT04337775
Title: The Reliability and Validity of the Turkish Version of the Smartphone Impact Scale
Brief Title: The Turkish Version of the Smartphone Impact Scale
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, MSc Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 3278
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2020-07

CONDITIONS: Addiction Psychological; Healthy; Addiction
Keywords: smartphone; technological addiction; smartphone psychosocial impact; smartphone use
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Smartphone Impact Scale (SIS) was originally developed in English to determine the cognitive, affective, social, and behavioral impacts of smartphones in everyday life. The purpose of this study was to translate and cross-culturally adapt the SIS instrument into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
Smartphone Impact Scale (SIS) was originally developed in English to determine the cognitive, affective, social, and behavioral impacts of smartphones in everyday life. The purpose of this study was to translate and cross-culturally adapt the SIS instrument into Turkish and investigate its psychometric properties. Two hundred healthy young adults will include. For cross-cultural adaptation, two bi-lingual translators used the back-translation procedure. Within a 5-to-7-day period after the first assessment, the participants completed the Turkish version of SIS (SIS-T) to evaluate test-retest reliability. Cronbach's alpha (α) was used to assess internal consistency. The correlations with the Turkish version of the Smartphone Addiction Scale (SAS-T) and Turkish version of the Nottingham Health Profile (NHP-T) will determine to check the validity.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35 years
* Having a smartphone that was connected to the Internet for at least 6 months
* Being a volunteer to participate

Exclusion Criteria:

* Having cognitive impairment
* Having disabilities in understanding, speaking and reading Turkish

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample will consist of volunteer, healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Smartphone Impact Scale | Baseline (First assessment)
  The Smartphone Impact Scale is a reliable and scale for evaluating cognitive, affective, social, and behavioral impacts of smartphones in everyday life. It assesses loss of control of smartphone use ,nomophobia, smartphone-mediated communication, emotion regulation through smartphone usage, smartphone support to romantic relationships, smartphone tasks support, and awareness of smartphone negative impact. A high score in the subscales shows a higher negative impact of smartphone on cognitive, affective, social, and behavioral aspects.

SECONDARY OUTCOMES:
Smartphone Impact Scale | Within a 5-to-7-day period after the first assessment (Second assessment)
  The Smartphone Impact Scale is a reliable and scale for evaluating cognitive, affective, social, and behavioral impacts of smartphones in everyday life. It assesses loss of control of smartphone use ,nomophobia, smartphone-mediated communication, emotion regulation through smartphone usage, smartphone support to romantic relationships, smartphone tasks support, and awareness of smartphone negative impact. A high score in the subscales shows a higher negative impact of smartphone on cognitive, affective, social, and behavioral aspects.
Smartphone Addiction Scale | Baseline (First assessment)
  Smartphone Addiction Scale (SAS) is a self-reported scale developed by Kwon et al. based on internet addiction and the features of smartphones in 20135. The scale consisted of 33 items rated on a 6-point Likert-type scale from 1 to 6. A high total score in the scale, which has no cut-off score, shows a smartphone addiction risk. The Turkish version of SAS (SAS-T), which was previously reported as a reliable instrument, will use in the present study.
Nottingham Health Profile | Baseline (First assessment)
  Nottingham Health Profile is patient-completed questionnaire used to determine and quantify perceived health problems. Composed of 38 items divided into six domains: 1) sleep, 2) mobility, 3) energy, 4) pain, 5) emotional reactions, 6) social isolation. Total Score ranges from 0 (no perceived distress) to 100 (maximum perceived distress). The Turkish version of Nottingham Health Profile, which was previously reported as a reliable and valid instrument, will use in the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya Mutlu, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

REFERENCES:
- [Derived] Birinci T, Van Der Veer P, Mutlu C, Mutlu EK. The Reliability and Validity of the Turkish Version of Smartphone Impact Scale. Eval Health Prof. 2023 Mar;46(1):84-91. doi: 10.1177/01632787221097703. Epub 2022 May 16. PMID 35575445